CLINICAL TRIAL: NCT05115825
Title: Survivors of Head and Neck Cancer: Optimizing Pain Management
Brief Title: Pain Management for Head and Neck Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: American Cancer Society, Inc. (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Shannon Madore, Ph.D., Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00019309; NCI-2021-10801 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00019309 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2021-10-29; First posted 2021-11-10 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Head and Neck Carcinoma
MeSH Terms: interventions — Behavior Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (Mobile Pain Coping Skills Training) (Experimental): Patients attend 5 sessions of Mobile Pain Coping Skills Training for 45 minutes each over 8 weeks.
  Interventions: Behavioral: Behavioral Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Attend Mobile Pain Coping Skills Training
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial improves an existing pain management program and tests its effect on head and neck cancer survivors. This trial aims to find a better program to improve pain-related physical functioning, mood, and quality of life in a sample of individuals who have undergone treatment for head and neck cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Adapt an existing telehealth pain management intervention to target improvement of pain-related physical functioning, mood, substance use, and quality of life in a local sample of veteran head and neck cancer (HNC) survivors.

II. Conduct a pilot of the adapted intervention to examine the feasibility (accrual, adherence, attrition) and acceptability (participant satisfaction) that will form the basis of a well-powered, randomized clinical trial submitted for funding to the National Institutes of Health (NIH), American Cancer Society (ACS), or Veterans Affairs (VA).

OUTLINE:

Patients attend 5 sessions of Mobile Pain Coping Skills Training for 45 minutes each over 8 weeks.

After completion of study, patients are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed diagnosis of HNC for which the participants have completed curative cancer treatment at the VA hospital or Oregon Health & Science University (OHSU) within the 3-12 months following treatment
* Self-reported current pain of 4 or higher, using the 0-10 Numeric Pain Rating (NRS) (0="no pain" to 10="the worst pain imaginable")
* Self-report of pain 4 or higher on two occasions, more than three weeks apart, since the completion of curative treatment

Exclusion Criteria:

* Enrolled in hospice
* Have substantial hearing or visual difficulties that would impair ability to participate
* Have inadequate cognitive functioning as indicated by medical record review and/or interactions with clinical staff. If needed the investigators can follow up with the St. Louis University Mental State Examination (score of < 22/30) (SLUMS); or
* Have untreated severe psychiatric illness that would impact the ability to consent and participate in the intervention
* Had only surgical treatment for their HNC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Pain-interference | Up to 2 months
  Will be assessed by Brief Pain Inventory. Will be assessed as 1-4=mild pain; 5-6 moderate pain; 7-10 severe pain.
Depression | Up to 2 months
  Will be assessed by the Patient Health Questionnaire. Scores of 5, 10, 15, and 20 represent point scale for mild, moderate, moderately severe and severe depression, respectively.
Pain coping self-efficacy | Up to 2 months
  Will be assessed by the Chronic Pain Self-Efficacy Scale.

SECONDARY OUTCOMES:
Substance use | Up to 2 months
  Will be assessed by the PENN Cravings Questionnaire. Total score >20 were considered to meet the threshold of craving, 15-20 were considered subthreshold, and <15 were considered non-cravers.
Head and neck cancer related quality of life | Up to 2 months
  Will be assessed by the University of Michigan Quality of Life Questionnaire.

OTHER OUTCOMES:
Prescription opioid dose | Up to 2 months
  Will be assessed via patient report.
Prescription opioid misuse | Up to 2 months
  Will be assessed using the Chronic Opioid Misuse Measure (COMM). A score of 9 or greater is suggestive of current problematic drug-related behaviors.
Patient acceptability | Up to 2 months
  Post-intervention, patients will be asked to rate satisfaction with the program, perception of utility with pain management, using a Likert-scale. Will inquire about patients' experiences participating in the intervention, perceived burden of participation, perception of the intervention utility, ease of use of the associated technology, and suggestions for improving the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shannon Madore, Ph.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (2):
- United States (2):
  - OHSU Knight Cancer Institute, Portland, Oregon
  - Portland VA Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Undecided